CLINICAL TRIAL: NCT06408584
Title: Short-course Hypofractionated Radiotherapy in Combination With Raltitrexed and Tislelizumab in Patients With Region-relapsed or Progressive Esophageal Squamous Cell Carcinoma: a Single Arm, Observational Study
Brief Title: Short-course Hypofractionated Radiotherapy in Combination With Raltitrexed and Tislelizumab
Acronym: SCHRT
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-ky117
Record Dates: First submitted 2024-03-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; tirelesizumab; Raltitrexed; Short course hypofractionated radiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study was to explore the safety and efficacy of short course hypofractionated radiotherapy combined with Raltitrexed and Tislelizumab in the treatment of patients with relapsed or advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signing informed consent; ECOG 0-2 points;
* Age over 18 years old, gender is not limited;
* Esophageal squamous cell carcinoma confirmed by pathology or clinically diagnosed by imaging;
* Recurrence of the tumor area after radical surgery or radical chemoradiotherapy; Regional progression of advanced esophageal squamous cell carcinoma after first-line or second-line treatment;
* Clinical staging: regional recurrence (rT0-4N0-3M0-1a) or regional progression (cT0-4N0-3M0-1) (AJCC/UICC esophageal cancer staging (8th edition));
* Tumor lesions can be evaluated;
* Expected survival ≥3 months;
* Major organ function is normal, meeting the following criteria: (i) blood routine examination A.HB ≥90g/L; b.ANC≥1.5×109/L; C. PLT ≥80×109/L; (ii) Biochemical examination: a. ALT/AST≤2.5ULN; b. TBIL≤1.5ULN; c. Plasma Cr≤1.5ULN or creatinine clearance (CCr)≥60ml/min;
* Women of childbearing age must have had a pregnancy within 7 days before starting treatment and the result is negative;
* All enrolled patients should take adequate contraceptive measures throughout the treatment period and 4 weeks after completion;
* no serious hematopoietic function, heart function, endocrine and immune function defects;
* No patients with grade 3 or above other serious medical diseases.

Exclusion Criteria:

* Under 18 years of age; ECOG is greater than 2;
* The diagnosis of esophageal cancer is not supported by pathological biopsy or image examination;
* Salvage surgery was performed after tumor recurrence;
* The patient has any active autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; The patient had vitiligo; Those with complete remission of asthma in childhood can be included without any intervention in adulthood; Patients with asthma requiring medical intervention with bronchodilators are not included);
* Patients who were taking immunosuppressants or systemic hormone therapy for immunosuppressive purposes (doses >10mg/ day of prednisone or other therapeutic hormones) and continued to use within 2 weeks before enrollment;
* Patients with severe and/or uncontrolled concomitant disease of grade 3 or higher, including: poor blood pressure control, myocardial ischemia or myocardial infarction, arrhythmia, active or uncontrolled severe infection; Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA≥104 copy numbers /ml or 2000IU/ml), or hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower detection limit of analytical methods);
* Pregnant or lactating women;
* Patients who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
* Patients who have participated in clinical trials of other drugs within four weeks; .Patients or family members refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with region-relapsed or progressive esophageal squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 month post treatment]
  progression free survival

SECONDARY OUTCOMES:
ORR | 1 month post treatment]
  objective response rate
1，3-year overall survival, Adverse effect | 1 month post treatment]
  overall survival, Adverse effect

CONTACTS AND LOCATIONS:
Locations (1):
- Yuan He, Hefei, China